CLINICAL TRIAL: NCT03367052
Title: Clinical and Radiological Outcomes of a 7-year Follow-up, Multi-center, Prospective, Randomized, Controlled Trial: Two-level Cervical ProDisc-C Vivo Versus Hybrid Construct.
Brief Title: Clinical and Radiological Outcomes: Two-level Cervical ProDisc-C Vivo Versus Hybrid Construct.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, guochen, Department of Spine Surgery, Peking University People's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: twolevelprodiscC
Record Dates: First submitted 2017-11-29; First posted 2017-12-08 (Actual); Last update posted 2017-12-08 (Actual); Status verified 2017-12

CONDITIONS: Cervical Disc Disease
Keywords: ProDisc-C vivo; Hybrid; Cervical degenerative disc disease

STUDY DESIGN:
Intervention Model Description: 542 DDD patients (age from 20 to 70) from several hospitals matching the inclusion criteria will be randomly assigned to two groups (271 patients in each group). One group will be treated with two level ProDisc-C vivo disc replacement. The other group will be treated with hybrid construct. Clinical outcomes and radiological analysis will be compared between the two groups at 1.5, 3, 6, 12, 24, 36, 60, and 84 months after the surgical treatments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Two level Prodisc-C vivo (Experimental): Two level Prodisc-C vivo cervical artificial disc replacement.
  Interventions: Procedure: Two level Prodisc-C vivo
- Hybrid (Active Comparator): This group of patients will be treated with hybrid construct, i.e., one level of Prodisc-C vivo and one level of anterior cervical discectomy fusion (ACDF).
  Interventions: Procedure: Hybrid

INTERVENTIONS:
Procedure: Two level Prodisc-C vivo — Two level of Prodisc-C vivo artificial disc replacement will be done in one group of patients.
  Arms: Two level Prodisc-C vivo
Procedure: Hybrid — The hybrid method will be used in one group of patients.
  Arms: Hybrid

SUMMARY:
The objective of this study is to investigate the clinical and radiological results of two-level cervical ProDisc-C vivo versus hybrid construct.

DETAILED DESCRIPTION:
This is a prospective, randomized, multicenter trial at 7 years of follow-up comparing two level ProDisc-C vivo artificial cervical disc replacement and hybrid construct, i.e., combining ACDF (Anterior cervical discectomy fusion) and ProDisc-C vivo to treat degenerative disc disease (DDD). 542 DDD patients (age from 20 to 70) from several hospitals matching the inclusion criteria will be randomly assigned to two groups (271 patients in each group). One group will be treated with two level ProDisc-C vivo disc replacement. The other group will be treated with hybrid construct. Clinical outcomes and radiological analysis will be done at 1.5, 3, 6, 12, 24, 36, 60, and 84 months after the surgical treatments.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of degenerative disc disease with radiculopathy or myeloradiculopathy at 2 contiguous levels from C-3 to C-7.
* The symptom is unresponsive to nonoperative treatment for at least 6 weeks.
* The patient demonstrates progressive symptoms calling for immediate surgery.

Exclusion Criteria:

* Any prior cervical spine surgery.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 542 (Estimated)
Dates: Start 2018-01-01 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Change of overall success rate | The overall success will be assessed at each time point (1.5, 3, 6, 12, 24, 36, 60, and 84 months after the surgical treatments).
  A patient's outcome was considered an overall success if all of the following conditions were met:1) postoperative (Neck Disability Index) NDI score improvement of at least a 15-point increase from preoperative score; 2) maintenance or improvement in neurological status; 3) disc height success; 4) no serious adverse event classified as implant associated or implant/surgical procedure associated; and 5) no additional surgical procedure classified as a "failure".

SECONDARY OUTCOMES:
Change of sagittal angular motion | The radiographs will be obtained at each study point (before surgery,1.5, 3, 6, 12, 24, 36, 60, and 84 months after the surgical treatments).
  Neutral anteroposterior and lateral radiographs and dynamic flexion-extension lateral radiographs.
Change of NDI Scores | The NDI scores will be assessed at each study point (before surgery,1.5, 3, 6, 12, 24, 36, 60, and 84 months after the surgical treatments).
  The neck disability index(NDI) questionnaire measures the level of pain and disability associated with various activities. The NDI is a 10-item, 50-point index that assesses different aspects of daily functioning in patients with neck pain. Each item is scored 0 to 5. The NDI score is a sum of the scores of the10-item. Clinical effects will be evaluated based on scores of the NDI. Higher values represent a better outcome.
Change of Arm and Neck pain | Neck and arm pain scores will be measured at each study point (before surgery,1.5, 3, 6, 12, 24, 36, 60, and 84 months after the surgical treatments).
  Neck and arm pain scores will be measured using a visual analogue scale (VAS) from "0' (no sensation) to '100"(the most intense pain imaginable) where 30 means "pain threshold".

CONTACTS AND LOCATIONS:
Overall Officials: chen guo, Master, Principal Investigator — Peking University People's Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zigler JE, Delamarter R, Murrey D, Spivak J, Janssen M. ProDisc-C and anterior cervical discectomy and fusion as surgical treatment for single-level cervical symptomatic degenerative disc disease: five-year results of a Food and Drug Administration study. Spine (Phila Pa 1976). 2013 Feb 1;38(3):203-9. doi: 10.1097/BRS.0b013e318278eb38. PMID 23080427
- [Background] Davis RJ, Kim KD, Hisey MS, Hoffman GA, Bae HW, Gaede SE, Rashbaum RF, Nunley PD, Peterson DL, Stokes JK. Cervical total disc replacement with the Mobi-C cervical artificial disc compared with anterior discectomy and fusion for treatment of 2-level symptomatic degenerative disc disease: a prospective, randomized, controlled multicenter clinical trial: clinical article. J Neurosurg Spine. 2013 Nov;19(5):532-45. doi: 10.3171/2013.6.SPINE12527. Epub 2013 Sep 6. PMID 24010901